CLINICAL TRIAL: NCT04608071
Title: Efficacy and Safety of a Modified Method for Blind Bedside Placement of Post-pyloric Feeding Tube：a Randomized Controlled Trial
Brief Title: A Modified Method for Blind Bedside Placement of Post-pyloric Feeding Tube.
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2020-273
Record Dates: First submitted 2020-10-27; First posted 2020-10-29 (Actual); Last update posted 2020-11-02 (Actual); Status verified 2020-04

CONDITIONS: Nutritional Support, Catheterization, Post-pyloric Feeding Tube, Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- M group: In M group, patients underwent modified post-pyloric feeding tube bedside placement
  Interventions: Procedure: A modified method for blind bedside placement of post-pyloric feeding tube.
- C group: In C group, patients underwent conventional Corpak protocol
  Interventions: Procedure: A modified method for blind bedside placement of post-pyloric feeding tube.
- EM group: In EM group, patients received standard electromagnetic guided tube placement.
  Interventions: Procedure: A modified method for blind bedside placement of post-pyloric feeding tube.

INTERVENTIONS:
Procedure: A modified method for blind bedside placement of post-pyloric feeding tube. — Modified post-pyloric feeding tube bedside catheterization as an optimized bedside blind post-pyloric tube placement, significantly shortened the time for passing pylorus without causing any severe adverse reactions.

SUMMARY:
To compare efficacy and safety of a new modified post-pyloric feeding tube bedside catheterization with Corpak 10-10-10 protocol and electromagnetic guided catheterization for treatment of patients with dysphagia and at high-risk of aspiration pneumonia. We conducted a single-center, single-blinded, and randomized controlled clinical trial. A total of 63 patients were treated with the non-gravity type CORFLO gastrointestinal feeding tube between 2017.1 and 2019.1 using different procedures: in the M group, patients underwent modified post-pyloric feeding tube bedside placement; in C group, patients underwent conventional Corpak protocol; in EM group, patients received standard electromagnetic guided tube placement.

ELIGIBILITY:
Inclusion Criteria:

* All patients had dysphagia that could not be alleviated within 48 hours
* High-risk status with aspiration pneumonia, including consciousness disorder caused by various diseases, severe dementia, bed rest, gastroesophageal reflux, hiccup, gastric retention, achalasia of pyloric.
* Can't receive nasogastric tube feeding.

Exclusion Criteria:

* The previous history of upper abdominal surgery.
* Gastroduodenal ulcer and esophagogastric varices;
* Severe sinusitis and nasal bone fracture;
* Patients with recent gastrointestinal bleeding, intestinal obstruction, ischemic bowel disease, and epistaxis;
* Patients with electromagnetically-guided catheterization should additionally exclude implantable cardiac defibrillator, implantable cardiac pacemaker or diaphragm pacemaker.

Ages: 18 Years to 90 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Sixty-three patients with dysphagia from Department of Rehabilitation, the Second Affiliated Hospital of Zhejiang University School on January 1, 2017 to January 1, 2019. All the patients included in this study were in accordance with the guide of diagnosis and treatment of swallowing disorders of diagnostic criteria.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-01-01 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
The success rate of NIT placement | 2019.10
  The successful catheterization was defined when the catheter tip was placed behind the pylorus.

SECONDARY OUTCOMES:
Operation time of tube insertion | 2019.10
  The time spent on the catheterization.

OTHER OUTCOMES:
The time for passing pylorus and the depth of insertion | 2019.10
  The time the catheterization passes through the pylorus.
Serious complications | 2019.10
  asphyxiation, hemoptysis, and exacerbation of aspiration pneumonia

CONTACTS AND LOCATIONS:
Overall Officials: Xiong Bing, M.M.D, Principal Investigator — Department of Rehabilitation, The Second Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, 310009, PR China.

IPD SHARING:
Plan to Share IPD: No